CLINICAL TRIAL: NCT04323982
Title: Comparison of Traditional Cataract Surgery and Traditional Surgery Combine Triamcinolone Staining of the Anterior Vitreous in Treating Congenital Cataracts
Brief Title: Comparison of Traditional Cataract Surgery and Traditional Surgery Combined Triamcinolone Staining
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2020-China-1
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Congenital Cataract
Keywords: congenital cataract, Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Cataract Surgery (Experimental): Traditional surgery combined triamcinolone staining of the anterior vitreous (TA)
  Interventions: Procedure: new surgical procedure
- Traditional Cataract Surgery (Active Comparator): For patients younger than 2 years of age: anterior continuous capsulorhexis + irrigation/aspiration + posterior capsulorhexis + anterior vitrectomy (ACCC+ I/A + PCCC + A-vit) For patients older than 2years of age: anterior continuous capsulorhexis + irrigation/aspiration + posterior capsulorhexis + primary intraocular lens implantation + anterior vitrectomy (ACCC+ I/A + PCCC + IOL + A-vit)
  Interventions: Procedure: traditional surgical procedure

INTERVENTIONS:
Procedure: new surgical procedure — （ACCC + I / A + PCCC + TA+ A-vit) or （ACCC + I / A + PCCC + IOL + TA + A-vit）
  Arms: New Cataract Surgery
Procedure: traditional surgical procedure — （ACCC + I / A + PCCC + A-vit) or （ACCC + I / A + PCCC + IOL + A-vit）
  Arms: Traditional Cataract Surgery

SUMMARY:
Previously, the investigators have developed a surgical technique to reduce inflammatory response after congenital cataract surgery. This prospective, randomized controlled study aims to compare the prognosis of traditional cataract surgery with traditional surgery combined triamcinolone staining of the anterior vitreous in treating congenital cataracts.

DETAILED DESCRIPTION:
Surgical technique for congenital cataract is now more and more mature, but many young patients still have obvious postoperative inflammatory response, which might cause visual axial opacification, posterior synechiae and secondary glaucoma. Triamcinolone is used in intraocular injection for its anti-inflammatory effect However, the application of Triamcinolone was reported to be associated with high intraocular pressure. It is necessary to evaluate the safety and effectiveness of using triamcinolone in congenital cataract surgery.

In this randomized clinical trial, children with equal degree of congenital cataract in both eyesare enrolled. Patients receive cataract surgery on both eyes on the same day. For each patient, one eye is randomly assigned to undergo traditional surgical procedure, while the fellow eye is undergoing new surgical procedure. The traditional surgical procedure include anterior continuous curvilinear capsulorhexis (ACCC), irrigation/aspiration (I/A), posterior continuous curvilinear capsulorhexis (PCCC), and anterior vitrectomy(A-VIT). Primary intraocular lens implantation (IOL) is performed in children older than age of two. The new surgical procedure is to combine triamcinolone staining of the anterior vitreous on the basis of the traditional surgical procedure. Investigators then compare the incidence of high intraocular pressure, visual axis opacification, uveitis, iris/pupil abnormality, and macular edema between two groups

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 months and 13 years
2. Uncomplicated bilateral same degree of congenital cataract (≥ 3 mm central dense opacity)
3. Informed consent signed by a parent or legal guardian

Exclusion Criteria:

1. Intraocular pressure >21 mmHg
2. Preterm birth (<28 weeks)
3. Presence of other ocular diseases (keratitis, keratoleukoma, aniridia, glaucoma, microcornea, persistent hyperplastic primary vitreous) or systemic disease (congenital heart disease, ischemic encephalopathy)
4. History of ocular trauma
5. Previous intraocular surgery

Ages: 3 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
incidence of high intraocular pressure | 5 years
  Determined with the Tono-pen.
incidence of visual axis opacification | 5 years
  Visual axis obscuration will be evaluated based on the retroillumination.
incidence of uveitis and iris/pupil abnormality | 5 years
  Uveitis and iris/pupil abnormality will be evaluated based on the slip lamp examination.

SECONDARY OUTCOMES:
Best corrected visual acuity | 5 years
  Determined with the Teller's acuity card, the Lea symbol visual acuity chart or the ETDRS chart according the patient's age.
Central corneal thickness | 5 years
  Determined with the pentacam.
Central macular thickness | 5 years
  Determined with the optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Weirong, MD, Study Chair — SunYat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Homepage of Zhongshan Ophthalmic Center — http://www.gzzoc.com/